CLINICAL TRIAL: NCT01218685
Title: Evaluation Aof Safety and Immunogenicity of Non-adjuvanted Pandemic Influenza A (H1N1) Vaccine in Chronic and or Immunocompromised Patients, Elderly and Pregnants, Produced by Butantan Institute
Brief Title: Evaluation of Pandemic Influenza A (H1N1) Vaccine in Chronic and or Immunocompromised Patients, Elderly and Pregnants
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Collaborators: University of Sao Paulo (Other); Insituto Adolfo Lutz (Unknown); Centro de Referencia e Treinamento em DST/AIDS (Unknown)
Responsible Party: Sponsor
Other Study IDs: BUTVAC-Influenza A (H1N1) 2.0
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Immunocompromised Patients; Safety of Pandemic Influenza A (H1N1)Vaccine; Immunogenicity of Pandemic Influenza A (H1N1)Vaccine
Keywords: Immunocompromised patients; Safety of pandemic influenza A (H1N1)vaccine; Immunogenicity of pandemic influenza A (H1N1)vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- Health adults
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- Health children
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- Pregnants
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- Elderly over 65 years old
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- HIV patients
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- Kidney transplant
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- Oncologic patients
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- Rheumatologic adult patients
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS
- Rheumatologic children patients
  Interventions: Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS

INTERVENTIONS:
Biological: Split inactivated A/California/7/2009 (H1N1) (NYMC X-179A) VIRUS — 1 full dose of 15 micrograms, IM, for volunteers 9 years of age or older; children 6 months to 2 years of age, half of the dose,IM, with 21 days interval; children 3 years old up to 8 years old, 1 full dose, IM, twice, with 21 days interval.

SUMMARY:
The objective of this study is to describe the safety and immunogenicity of a non-adjuvanted vaccine against pandemic influenza A (H1N1)in patients with chronic and or immunocompromised disease, elderly and pregnants. The primary immunological endpoint is to analyze the proportion of subjects with antibody titers of 1:40 or more on hemagglutination-inhibition assay 21 days after 1 dose of the vaccine. Volunteers will be monitored for safety during 21 days after vaccination. Volunteers will be recruited based on inclusion and exclusion criteria. Vaccine composition is: 15 micrograms of split inactivated virus (A/California/7/2009 (H1N1) (NYMC X179A). The hypothesis of the study is that the vaccine is safe and immunogenic in the volunteers recruited.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers able to understand and agree to participate in the study.

Exclusion Criteria:

* Have egg allergy
* Have past history of allergy to seasonal influenza vaccine
* Have received another inactivated vaccine within the prior 2 weeks or live vaccine in the past four weeks to his/her participation in the study
* Acute infectious disease during seven days prior vaccination
* Confirmed prior infection by pandemic influenza A (H1N1)
* Have participated in another clinical trial in the last 6 months
* Any other condition identified by the principal investigators which is considered not safe for enrollment of the volunteer.

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers with chronic and or immunocompromised disease, elderly and pregnant in follow - up at the institutions participants in the study will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1152 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Antibody titers of 1:40 or more for influenza A pandemic (H1N1) | 21 days after vaccination
  the proportion of subjects with antibody titers of 1:40 or more on hemagglutination-inhibition assay

SECONDARY OUTCOMES:
Safety of the vaccine | 21 days after vaccination
  Evaluation of local and systemic adverse effects through the study period including 30 minutes after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Roberto Precioso, MD, PhD, Study Chair — Butantan Foundation
Locations (1):
- Avenida Vital Brasil 1500, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Miraglia JL, Abdala E, Hoff PM, Luiz AM, Oliveira DS, Saad CG, Laurindo IM, Viso AT, Tayra A, Pierrotti LC, Azevedo LS, Campos LM, Aikawa NE, Timenetsky Mdo C, Luna E, Cardoso MR, Guedes Jda S, Raw I, Kalil J, Precioso AR. Immunogenicity and reactogenicity of 2009 influenza A (H1N1) inactivated monovalent non-adjuvanted vaccine in elderly and immunocompromised patients. PLoS One. 2011;6(11):e27214. doi: 10.1371/journal.pone.0027214. Epub 2011 Nov 8. PMID 22087267